CLINICAL TRIAL: NCT02137109
Title: Meta-Analysis of the Safety and Efficacy of Natalizumab in Pediatric Patients With Multiple Sclerosis
Brief Title: Safety and Efficacy in Pediatric MS Patients Prescribed Tysabri
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 101MS028
Record Dates: First submitted 2014-05-01; First posted 2014-05-13 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Multiple Sclerosis
Keywords: Pediatric
MeSH Terms: conditions — Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- natalizumab: Natalizumab will not be provided as a part of this study. Participants will receive natalizumab per the local label specifications.
  Interventions: Drug: natalizumab

INTERVENTIONS:
Drug: natalizumab — Administered as specified in the treatment arm.
  Other Names: BG00002; Tysabri

SUMMARY:
The primary objective of the study is to evaluate the safety of natalizumab use in the pediatric multiple sclerosis (MS) population.

DETAILED DESCRIPTION:
All available retrospective and prospective data from pediatric MS participants who have received at least 1 dose of natalizumab before turning 18 years old and before 31Mar2015 will be used in this study. Prospective data are defined as data to be collected in the future, i.e., from new participants not included in the first data transfer or additional data from existing participants that were not included in the first data transfer. Existing biospecimen samples will be evaluated but not collected as part of this study.

ELIGIBILITY:
Key Inclusion Criteria:

* All available retrospective and prospective data from pediatric MS patients who have received at least 1 dose of natalizumab before turning 18 years old and before 31 March 2015.
* In addition, patients must be registered in TOUCH (US patients only), enrolled in a Biogen sponsored postmarketing observational study (e.g., TOP (NCT00493298) or TYGRIS (NCT00477113,NCT00483847)), or in a country-specific TYSABRI registry.
* Adequate data received by Biogen by 30 September 2015 will be used for this meta-analysis including data collected after a patient may have turned 18 years old.

Key Exclusion Criteria:

* Data received by Biogen after 30 September 2015 will not be included in the statistical analyses

NOTE: Other protocol-defined inclusion/exclusion Criteria May Apply

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric MS patients who have received at least 1 dose of natalizumab prior to the age of 18 years where the first dose was administered prior to 31 March 2015.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Incidence of all serious adverse events (SAEs) | Up to 19 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen